CLINICAL TRIAL: NCT03558230
Title: Sensory Stimulation During Constraint-Induced Movement Therapy
Brief Title: Sensory Stimulation During CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO74164
Record Dates: First submitted 2018-05-07; First posted 2018-06-15 (Actual); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy
Keywords: pediatric; hemiplegic; hand function
MeSH Terms: conditions — Cerebral Palsy | interventions — Vibration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blinded stratified randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration (Experimental): The experimental group will receive the wrist stimulation during standardized Constraint-Induced Movement Therapy.
  Interventions: Behavioral: Standardized Constraint-Induced Movement Therapy; Behavioral: Vibration
- No Vibration (Placebo Comparator): The control group will wear the vibration device with no vibration during standardized Constraint-Induced Movement Therapy.
  * The vibration device is a generic, commercially-available, vibrator, not particularly used for this peripheral skin stimulation purpose.
  Interventions: Behavioral: Standardized Constraint-Induced Movement Therapy; Behavioral: Placebo (for vibration)

INTERVENTIONS:
Behavioral: Standardized Constraint-Induced Movement Therapy — The standardized Constraint-Induced Movement Therapy aims to improve the child's weak upper extremity through intensive frequent and repetitive movements. The therapy duration is 6 hours/day for 5 consecutive days.
Behavioral: Vibration — Vibration applied to the wrist.
  Arms: Vibration
Behavioral: Placebo (for vibration) — No vibration applied to the wrist.
  Arms: No Vibration

SUMMARY:
The long-term goal of this project is to assess the impact of the novel sensory stimulation technique in enhancing outcomes of constraint-induced movement therapy (CIMT) in children with cerebral palsy. This is a pilot project.

DETAILED DESCRIPTION:
The stimulation is peripheral sensory stimulation involving application of low-level, random-frequency vibration to the wrist skin. The hypothesis is that improvement in upper extremity function will be greater for the experimental group receiving the stimulation during CIMT compared with the control group who will wear the device with no vibration (placebo). This pilot study is to assess feasibility and safety.

ELIGIBILITY:
* Between the ages of 3 and 9
* Have unilateral upper limb motor weakness.
* Use the affected extremity as a gross assist during play and self-care activities.
* No significant developmental delays that would limit spontaneous use of the more affected extremity.
* Be ambulatory for their age and demonstrate intact balance and protective reactions throughout the less involved upper extremity.
* No other health impairment other than hemiparesis.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2018-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Na Jin Seo, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vibration: The experimental group will receive the wrist stimulation during standardized Constraint-Induced Movement Therapy.
  Standardized Constraint-Induced Movement Therapy: The standardized Constraint-Induced Movement Therapy aims to improve the child's weak upper extremity through intensive frequent and repetitive movements. The therapy duration is 6 hours/day for 5 consecutive days.
  Vibration: Vibration applied to the wrist.
  The vibration device is a generic, commercially-available, vibrator, not particularly used for this peripheral skin stimulation purpose.
- No Vibration: The control group will wear the vibration device with no vibration during standardized Constraint-Induced Movement Therapy.
  Standardized Constraint-Induced Movement Therapy: The standardized Constraint-Induced Movement Therapy aims to improve the child's weak upper extremity through intensive frequent and repetitive movements. The therapy duration is 6 hours/day for 5 consecutive days.
  Placebo (for vibration): No vibration applied to the wrist.
  The vibration device is a generic, commercially-available, vibrator, not particularly used for this peripheral skin stimulation purpose.
Period: Overall Study
Arm/Group | Vibration | No Vibration
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibration | No Vibration | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.7 (1.8) | 5.5 (1.9) | 5.6 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 3 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Total Number of Hours That Participants Wear the Device)
Description: total number of hours that participants wear the device
Time Frame: through 5-day study completion.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vibration | No Vibration
Number analyzed (Participants) | 7 | 6
Hours | 28.3 (0.3) | 27.9 (1)

ADVERSE EVENTS:
Time Frame: Throughout the 5-day study period
Arm/Group | Vibration | No Vibration
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 2/7 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibration (N=7) | No Vibration (N=6)
Temporary skin redness (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03558230/Prot_SAP_000.pdf